CLINICAL TRIAL: NCT04644159
Title: Longitudinal Follow-up of a Population Cohort in a French City With High SARS-CoV-2 Circulation in Early 2020
Brief Title: Longitudinal Follow-up of a Population Cohort in a French City With High SARS-CoV-2 Circulation, in Early 2020 [COVID-19]
Acronym: COVID-OISE
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-060
Record Dates: First submitted 2020-11-18; First posted 2020-11-25 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: SARS (Severe Acute Respiratory Syndrome); Covid19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva, nasopharyngeal mucosa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Housolds: Pupils, teachers and non-teaching staff who attended schools of the city during the 2019-2020 school year and members of their households
  Interventions: Other: Human biological samples
- Subjects hospitalized or residing in health care facilities: Residents and patients from retirement homes and long-term care units
  Interventions: Other: Human biological samples
- Staff of health care institutions: Staff of health care institutions
  Interventions: Other: Human biological samples

INTERVENTIONS:
Other: Human biological samples — Blood , saliva, nasopharyngeal mucosa

SUMMARY:
An initial retrospective epidemiological investigation was conducted in a city north of France after the diagnosis of the first case of COVID-19 on February 2020. Sero-epidemiological studies were conducted in this town by the Institut Pasteur in early 2020 among families, teachers and non-teaching staff of the high and elementary schools.

The goal of this new project is to better characterize the specific immunity generated by the infection within this community. The specific immune response to the SARS-CoV-2 virus will be followed for a period of 2 years from the initial circulation of the virus, within a large cohort of participants covering all age groups from 5 years-old onwards. The study will focus on systemic humoral and cell responses, immunity of the nasopharyngeal mucosa and the humoral response present in saliva. Follow-up of participants in this cohort and monitoring of the virus circulation within this community would help to determine the protective character against re-infection of the natural immunity generated by SARS-CoV-2.

DETAILED DESCRIPTION:
An initial retrospective epidemiological investigation was conducted in a city north of France after the diagnosis of the first case of COVID-19 on February 2020. Sero-epidemiological studies were conducted in this town by the Institut Pasteur in early 2020 among families, teachers and non-teaching staff of the high and elementary schools.

These surveys have documented the circulation of SARS-CoV-2 in one of the first French COVID-19 outbreaks and this study proposes to better characterize the specific immunity generated by the infection among this community. Indeed, the nature of this immunity and its persistence over time are crucial information. The goal of this new project is to explore the specific immune response to the SARS CoV 2 virus for a period of 2 years from the initial circulation of the virus in this north of France city, within a large cohort of participants in the general population covering all age groups from 5 years of age but also in patients and residents of retirement homes in this city. It is expected that the immune response conferred by natural infection or vaccination will differ according to age.

This study will focus on systemic humoral and cell responses, immunity of the nasopharyngeal mucosa and the humoral response present in saliva. The genetic basis of the diversity of humoral responses induced by SARS-CoV-2 and those related to the multiplicity of clinical manifestations of COVID-19 will also be investigated. This would provide initial evidence to determine the protective character against re-infection of the natural immunity generated by CoV-2-SARS. Finally, these data will be used to model the intra-family transmission of the virus.

ELIGIBILITY:
Inclusion Criteria:

* Adultes and minors from 5 years old
* Affiliated with or benefiting from a Social Security system
* State of health compatible with a blood sample as defined in the protocol

Exclusion Criteria:

* Person benefiting from a legal protection measure or unable to express informed consent to participation and for which the legal representative or tutor person could not be contacted.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pupils, their parents and siblings, as well as teachers and non-teaching staff of a high and elementary schools located in a city north of France.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Presence of specific anti-SARS-CoV-2 antibodies in the different study groups. | 2 years
  Description of the serological status of individuals

SECONDARY OUTCOMES:
Presence of specific T cell response to the SARS-CoV-2 | 2 years
  Detection over time the specific T cell response to the SARS-CoV-2 virus.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Noëlle Ungeheuer, Dr, Principal Investigator — Institut Pasteur
Locations (2):
- France (2):
  - Hôpital de Crépy en Valois, Crépy-en-Valois
  - Institut Pasteur, Paris

IPD SHARING:
Plan to Share IPD: Undecided